CLINICAL TRIAL: NCT06591091
Title: Clemastine for Improving White Matter and Boosting Antidepressant Response in Late-life Depression
Acronym: CLIMB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, Olusola Alade Ajilore, Professor. Director, Clinical Research Core/Center for Clinical and Translational Science, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0636
Record Dates: First submitted 2024-08-05; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Depression
Keywords: Late-life Depression; Antidepressant medication response
MeSH Terms: conditions — Depression | interventions — Clemastine

STUDY DESIGN:
Intervention Model Description: The design of this pilot study is a randomized double-blind, placebo-controlled design with one arm standard antidepressant treatment plus placebo (n=20) and one arm standard antidepressant treatment plus clemastine (5.36 mg PO daily; n=60) for 12 weeks with primary outcomes related to improvement in the level of depression and white matter integrity.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The design of this pilot study is a randomized double-blind. Only the study Pharmacist will be unblinded to the placebo-controlled design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clemastine arm (Experimental): Participants in the clemastine arm of the study will receive clemastine 5.36 mg PO twice daily for 12 weeks. Based on clinical assessment, participants will also receive one of the following antidepressant medications: SSRI: Fluoxetine, sertraline, citalopram, escitalopram, vilazodone, vortioxetine SNRI: Venlafaxine, desvenlafaxine, duloxetine, levomilnacipran Augmentation: Bupropion and mirtazapine (monotherapy option in addition to first augmentation level), aripiprazole and quetiapine (second augmentation level).
  Allowable concomitant medications parallel clinical practice. These can include trazodone (up to 100mg nightly) for insomnia or as-needed use of benzodiazepines for concomitant anxiety, up to a maximum daily dose equivalent to lorazepam 2mg daily. Psychotropic medications used for other indications (such as tricyclics or gabapentin for pain) are allowable. Concomitant psychotherapy is allowed.
  Interventions: Drug: Clemastine Fumarate
- Placebo arm (Placebo Comparator): Participants in the placebo arm of the study will receive a placebo capsule PO twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clemastine Fumarate — Listed in arm/group description
  Other Names: Clemastine; Tavist Allergy
  Arms: Clemastine arm
Drug: Placebo — Listed in arm/group description
  Arms: Placebo arm

SUMMARY:
The goal of this study is to find out if the antihistamine, clemastine, can make the white matter in the brain better in older adults with depression. The study will also determine whether this improvement can make antidepressant treatment work better, reduce depressive symptoms, and improve memory and thinking.

DETAILED DESCRIPTION:
Geriatric depression, also known as late-life depression, is a type of major depression that affects people who are 60 years old or older. It can be difficult to treat and often comes back after treatment. It can also lead to problems with memory and thinking. Some studies have found that problems with the white matter in the brain can make it harder to treat depression in older adults. White matter helps with communication in the brain. A new study suggests that a medicine called clemastine might be able to improve the white matter in the brain. Clemastine is usually used as an antihistamine, but it might also help the brain repair itself. The goal of this study is to find out if clemastine can make the white matter in the brain better in older adults with depression. The study will also determine whether this improvement can make antidepressant treatment work better, reduce depressive symptoms, and improve memory and thinking. The study will involve two groups of participants. One group will receive the standard antidepressant treatment along with a placebo, while the other group will receive the standard antidepressant treatment along with clemastine. The investigators will compare the effects of these two treatments over a period of 12 weeks. The investigators will measure the improvement in white matter using special brain imaging techniques. The investigators will also assess the participants' mood, memory, and thinking abilities, and keep track of any side effects or problems caused by the treatments. Overall, this study has the potential to contribute valuable insights into the treatment of geriatric depression, alleviate depressive symptoms, enhance cognitive function, and potentially open up new avenues for future research and therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Diagnosis of major depressive disorder, single or recurrent episode (DSM5)
* Symptom Severity: MADRS ≥ 15
* Seeking antidepressant treatment
* Cognition score of MoCA >24
* Fluent in English or Spanish

Exclusion Criteria:

* Other Axis I psychiatric disorders, except for simple phobia or anxiety disorders present uniquely during the depressive episode (e.g., generalized anxiety disorder (GAD) or panic disorder symptoms)
* History of alcohol or drug dependence or abuse in the last year
* History of a developmental disorder or history of IQ (intelligence quotient) <70
* Acute suicidality ideation within the past month as determined by the Columbia Suicide Severity Rating Scale (C-SSRS)
* Acute grief (<1 month)
* Current or past psychosis
* Primary neurological disorder, including dementia, clinical stroke, brain tumor, epilepsy, etc.
* Presence of unstable medical illness requiring urgent treatment
* Any MRI contraindication
* Electroconvulsive Therapy (ECT) in last 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Frequency, Intensity and Burden of Side Effects Rating Scale | 12 weeks
  The investigator will examine the safety of clemastine using the Frequency, Intensity, and Burden of Side Effects Rating Scale (FIBSER).
  The FIBSER is scored from 0-6, with higher scores indicating worse outcomes
Montgomery-Asberg Rating Scale for Depression | 12 weeks
  The investigators will examine the effectiveness of an antidepressant plus clemastine (5.36 mg twice daily) compared to antidepressant plus placebo on clinical outcomes as indexed by the Montgomery-Asberg Rating Scale for Depression (MADRS).
  The MADRS is scored from 0-60, with higher scores indicating a worse outcome
Quantitative Anisotropy | 12 weeks
  The investigators will measure the impact of an antidepressant plus clemastine (5.36 mg twice daily) compared to antidepressant plus placebo on white matter integrity as indexed by change in quantitative anisotropy (QA).
  QA has no units but is measured from 0 to 1 and a higher indicates better white matter integrity
Fractional Anisotropy | 12 weeks
  The investigators will measure the impact of an antidepressant plus clemastine (5.36 mg twice daily) compared to antidepressant plus placebo on white matter integrity as indexed by change in fractional anisotropy (FA).
  FA has no units but is measured from 0 to 1 and a higher indicates better white matter integrity

SECONDARY OUTCOMES:
Trail Making Test Part A and Part B | 12 weeks
  The investigators will examine the effectiveness of an antidepressant plus clemastine (5.36 mg twice daily) compared to antidepressant plus placebo on cognitive outcomes as indexed by Trail Making Test Parts A and B.
  The Trail Making Test A and B is scored by the time to completion (seconds) and number of errors, with higher scores indicating worse performance.
  For TMT Part A and Part B, the "average" and "deficient" scores are categorized as follows:
  TMT Part A 29 seconds (average) Over 79 seconds (Deficient) TMT Part B 75 seconds (average) Over 273 seconds (Deficient)
Orientation Dispersion Index | 12 weeks
  The investigators will measure the impact of an antidepressant plus clemastine (5.36 mg twice daily) compared to antidepressant plus placebo on white matter integrity as indexed by change in neurite orientation dispersion and density imaging (NODDI)-derived orientation dispersion index (ODI).
  The ODI has no units but ranges from 0-1, with higher values indicating more neurite dispersion.
Neurite Density Index | 12 weeks
  The investigators will measure the impact of an antidepressant plus clemastine (5.36 mg twice daily) compared to antidepressant plus placebo on white matter integrity as indexed by change in neurite orientation dispersion and density imaging (NODDI)-derived measured neurite density index (NDI).
  The NDI has no units but ranges from 0-1, with higher values indicating more intracellular diffusion

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data will made available upon request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be available approximately one year after the study is completed and will be available for the duration specified by the Sponsor.

REFERENCES:
- [Background] Green AJ, Gelfand JM, Cree BA, Bevan C, Boscardin WJ, Mei F, Inman J, Arnow S, Devereux M, Abounasr A, Nobuta H, Zhu A, Friessen M, Gerona R, von Budingen HC, Henry RG, Hauser SL, Chan JR. Clemastine fumarate as a remyelinating therapy for multiple sclerosis (ReBUILD): a randomised, controlled, double-blind, crossover trial. Lancet. 2017 Dec 2;390(10111):2481-2489. doi: 10.1016/S0140-6736(17)32346-2. Epub 2017 Oct 10. PMID 29029896
- [Background] Caverzasi E, Papinutto N, Cordano C, Kirkish G, Gundel TJ, Zhu A, Akula AV, Boscardin WJ, Neeb H, Henry RG, Chan JR, Green AJ. MWF of the corpus callosum is a robust measure of remyelination: Results from the ReBUILD trial. Proc Natl Acad Sci U S A. 2023 May 16;120(20):e2217635120. doi: 10.1073/pnas.2217635120. Epub 2023 May 8. PMID 37155847
- [Background] Marawi T, Ainsworth NJ, Zhukovsky P, Rashidi-Ranjbar N, Rajji TK, Tartaglia MC, Voineskos AN, Mulsant BH. Brain-cognition relationships in late-life depression: a systematic review of structural magnetic resonance imaging studies. Transl Psychiatry. 2023 Aug 19;13(1):284. doi: 10.1038/s41398-023-02584-2. PMID 37598228